CLINICAL TRIAL: NCT05918328
Title: A Non Inferior, Randomized Controlled Phase II Clinical Study Comparing the Efficacy of Nab-PH+Pyrrolitinib and TCbHP in the Neoadjuvant Treatment of HER2 Positive Breast Cancer
Brief Title: Comparing the Efficacy of Nab-PH+Pyrrolitinib and TCbHP in the Neoadjuvant Treatment of HER2 Positive BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-013
Record Dates: First submitted 2023-06-11; First posted 2023-06-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; pathologic complete response; Pyrrolitinib; Disease-free survival
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria were randomly divided into TCbHP group and Nab-PH+pyrrolitinib group in a 1:1 ratio.
Masking Description: Non
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-PH+pyrrolitinib regimen group (Experimental): Drug dose of Nab PH+pyrrolitinib scheme: albumin paclitaxel （260mg/㎡ every 3 weeks or 125mg/㎡ weekly）+trastuzumab (initial loading dose 8 mg/kg, sequential maintenance dose 6 mg/kg, once every 3 weeks)+pyrrolitinib (320mg, QD), 3 weeks as one cycle.
  Interventions: Drug: Albumin paclitaxel+trastuzumab+pyrrolitinib
- TCbHP regimen group (Placebo Comparator): The drug dose of TCbHP protocol: docetaxel 75 mg/m2+carboplatin (AUC=6)+trastuzumab (initial load dose 8 mg/kg, sequential maintenance dose 6 mg/kg)+patuzumab (initial load dose 840mg, sequential maintenance dose 420 mg), one cycle every 21 days.
  Interventions: Drug: Docetaxel+Carboplatin+trastuzumab+Parstuzumab

INTERVENTIONS:
Drug: Albumin paclitaxel+trastuzumab+pyrrolitinib — albumin paclitaxel （260mg/㎡ every 3 weeks or 125mg/㎡ weekly）+trastuzumab (initial loading dose 8 mg/kg, sequential maintenance dose 6 mg/kg, once every 3 weeks)+pyrrolitinib (320mg, QD), 3 weeks as one cycle.
  Other Names: Nab-PH+pyrrolitinib regimen
  Arms: Nab-PH+pyrrolitinib regimen group
Drug: Docetaxel+Carboplatin+trastuzumab+Parstuzumab — Docetaxel 75 mg/m2+carboplatin (AUC=6)+trastuzumab (initial loading dose 8 mg/kg, sequential maintenance dose 6 mg/kg)+patuzumab (initial loading dose 840mg, sequential maintenance dose 420 mg), one cycle every 21 days
  Other Names: TCbHP regimen
  Arms: TCbHP regimen group

SUMMARY:
At present, the incidence rate of breast cancer has exceeded that of lung cancer, becoming the largest cancer in the world. HER2 overexpression breast cancer accounts for about 20%~30% of all breast cancer patients. HER2 is an important prognostic indicator and therapeutic target for breast cancer. Targeted therapy for HER2 protein is the core treatment of this type of breast cancer. Previous studies have confirmed that TKI drugs can reverse the resistance of large molecule monoclonal antibodies to a certain extent; Moreover, due to the complementarity of therapeutic targets, monoclonal antibodies are associated with TKI Drugs have synergistic effects. TCbHP is one of the preferred neoadjuvant chemotherapy schemes recommended by NCCN guidelines for HER2 positive breast cancer, but its incidence of adverse reactions such as vomiting, diarrhea, anemia, thrombocytopenia is significantly higher than that of the scheme without platinum. In the GeparOcto study and Geparsixto study, based on anthracycline+purple shirt+double target, the addition of carboplatin did not further improve the PCR rate of HER2 positive breast cancer neoadjuvant therapy. GeparSepto research showed that compared to the solvent based paclitaxel group, albumin paclitaxel increased the pCR rate by 8.2% and the IDFS by 7.3%. In the CA024 study, compared to docetaxel, albumin paclitaxel also significantly increased ORR and PFS. In the study by Lavasani SM et al., the neoadjuvant therapy of albumin paclitaxel combined with topiramate achieved a PCR rate of 64%. Therefore, we assume that the new adjuvant treatment scheme of Nab PH+pyrrolitinib can not be inferior to the efficacy of TCbHP, and has a lower incidence of adverse reactions, which may become a new adjuvant treatment option for HER2 positive breast cancer patients.

DETAILED DESCRIPTION:
At present, the incidence rate of breast cancer has exceeded that of lung cancer, becoming the largest cancer in the world. HER2 overexpression breast cancer accounts for about 20%~30% of all breast cancer patients. HER2 is an important prognostic indicator and therapeutic target for breast cancer. Targeted therapy for HER2 protein is the core treatment of this type of breast cancer. Previous studies have confirmed that TKI drugs can reverse the resistance of large molecule monoclonal antibodies to a certain extent; Moreover, due to the complementarity of therapeutic targets, monoclonal antibodies are associated with TKI Drugs have synergistic effects. TCbHP is one of the preferred neoadjuvant chemotherapy schemes recommended by NCCN guidelines for HER2 positive breast cancer, but its incidence of adverse reactions such as vomiting, diarrhea, anemia, thrombocytopenia is significantly higher than that of the scheme without platinum. In the GeparOcto study and Geparsixto study, based on anthracycline+purple shirt+double target, the addition of carboplatin did not further improve the PCR rate of HER2 positive breast cancer neoadjuvant therapy. GeparSepto research showed that compared to the solvent based paclitaxel group, albumin paclitaxel increased the pCR rate by 8.2% and the IDFS by 7.3%. In the CA024 study, compared to docetaxel, albumin paclitaxel also significantly increased ORR and PFS. In the study by Lavasani SM et al., the neoadjuvant therapy of albumin paclitaxel combined with topiramate achieved a PCR rate of 64%. Therefore, we assume that the new adjuvant treatment scheme of Nab PH+pyrrolitinib can not be inferior to the efficacy of TCbHP, and has a lower incidence of adverse reactions, which may become a new adjuvant treatment option for HER2 positive breast cancer patients. This study aims to explore the efficacy and safety of TCbHP * 6 and Nab-PH+pyrrolitinib * 6 as two new adjuvant treatment regimens in HER2 positive patients through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old, ECOG 0-1 point.
2. Clinical T2-T4d, or T1c with axillary LN+.
3. HER2+, invasive breast cancer confirmed by histopathology;(HER2 positive expression means that there is at least one case of tumor cell immunohistochemical staining intensity of 3+or positive confirmed by fluorescence in situ hybridization [FISH] in the pathological test/review of the primary focus conducted by the Pathology Department of the Research Center Hospital).
4. Having clinically measurable lesions: measurable lesions displayed on ultrasound, mammography, or MR (optional) within the first month of randomization.
5. Organ and bone marrow function tests within one month before chemotherapy indicate no contraindications to chemotherapy:Absolute value of neutrophil count ≥ 2.0 × 109/L; Hemoglobin ≥ 90g/L; Platelet count ≥ 100 × 109/L;Total bilirubin<1.5 ULN (upper limit of normal value); Creatinine<1.5 × ULN; AST/ALT < 1.5 × ULN.
6. Cardiac ultrasound: Left ventricular ejection fraction (LVEF ≥ 55%).
7. Women of childbearing age tested negative for serum pregnancy test 14 days before randomization.
8. Sign an informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. Has received chemotherapy, endocrine therapy, targeted therapy, reflex therapy, etc. for this disease.
3. The patient has a second primary malignant tumor, except for fully treated skin cancer.
4. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical procedures.
5. Serious heart disease or discomfort, including but not limited to the following diseases:Confirmed history of heart failure or systolic dysfunction (LVEF<50%); High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate>100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block; Angina pectoris requiring treatment with anti angina drugs; Clinically significant heart valve disease; ECG shows transmural myocardial infarction; Poor control of hypertension (systolic blood pressure>180 mmHg and/or diastolic blood pressure>100 mmHg).
6. Due to serious and uncontrollable other medical diseases, researchers believe that there are contraindications to chemotherapy.
7. Individuals with a known history of allergies to the drug components of this protocol; Having a history of immunodeficiency, including HIV testing positive, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR rate) | immediately after the intervention
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years after surgery
  EFS was defined as the time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or death from any cause.
DFS | 5-10 years after surgery
  Disease-free Survival,From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
Distant Disease Free Survival (DDFS) | 5-10 years after surgery
  DDFS is defined as the time from surgery to distant recurrence or death from any cause
Objective Response Rate (ORR) | Preoperative
  ORR is defined as the number of target lesion responders as assessed by MRI
number of adverse events | during each cycle of chemotherapy (21 days as 1 cycle)
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

OTHER OUTCOMES:
Multiple gene testing | immediately after surgery
  Exploring Multiple Gene Prediction Models for PCR Influencing Different Neoadjuvant Therapy Schemes

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Study Principal Investigator
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China